CLINICAL TRIAL: NCT06092320
Title: Outcome of a Lecture Before vs After Simulation-based Education on Pediatric Status Epileptics: A Randomized Controlled Pilot Trial
Brief Title: Does Teaching Before or After Simulation Improve Learning?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Melissa Chan, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H22-03760
Record Dates: First submitted 2023-10-03; First posted 2023-10-23 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Medical Education; Simulation
Keywords: Medical Education; Simulation; Pediatrics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know the specific pediatric resuscitation simulation they will be completing.
  Simulation reviewers will not know which arm of the intervention the participants are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation - Didactic Lecture Group (Experimental): This group will start with a Simulation and debrief followed by a didactic lecture afterwards. They will then complete a simulation 2 months later.
  Interventions: Other: Simulation on Pediatric Status Epilepticus; Other: Didactic Lecture on Pediatric Status Epilepticus
- Didactic Lecture - Simulation Group (Experimental): This group will start with a didactic lecture and then complete a simulation and debrief. They will then complete a simulation 2 months later.
  Interventions: Other: Simulation on Pediatric Status Epilepticus; Other: Didactic Lecture on Pediatric Status Epilepticus

INTERVENTIONS:
Other: Simulation on Pediatric Status Epilepticus — The participants will complete a simulation session and debrief lead by a pediatric emergency medicine physician on status epilepticus.
Other: Didactic Lecture on Pediatric Status Epilepticus — The participants will complete a lecture on pediatric status epilepticus

SUMMARY:
The goal of the randomized educational intervention study is to test whether simulation preceding didactic teaching leads to improved knowledge and performance retention compared to a didactic lecture proceeding simulation for medical students

Participants will be randomized to one of two different groups with reverse orders for simulation and lectures.

Researchers will compare each group to see which way is better for learning.

ELIGIBILITY:
Inclusion Criteria:

- Second year medical student at the University of British Columbia

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in resuscitation performance retention score 2 months post-initial training assessed using global simulation performance score | From initial simulation until repeat simulation 2 months later
  The scoring sheet used will be the Global Simulation performance score a one to seven scale that assess over medical expertise performance in the simulation with higher values representing increased competence.

SECONDARY OUTCOMES:
Change in knowledge assessment score at 2 months post-initial training assessed using an MCQ | From initial knowledge test until repeat testing 2 months later
  The knowledge test is a 15 questions multiple choice exam scored from 0 to 15 with higher numbers representing a higher score.
Learner satisfaction measured by Likert scale items after each simulation debrief | Single time metric completed five minutes after initial simulation session
  The Likert scale will be a one to five scale with higher scores representing increased satisfaction
Time to resuscitation metrics | The time for each metric will be measured once during the second evaluatory simulation 2 months after the initial simulation and participant enrolment.
  The following "time to" metrics will be measured from simulation start until completion of each activity within that simulation: glucose check, IV access, first-line anti-epileptic administration, second-line anti-epileptic administration, chemistry panel

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Chan, MD, Principal Investigator — Provincial Health Services Authority British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT06092320/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT06092320/ICF_001.pdf